CLINICAL TRIAL: NCT00133289
Title: Ventricular Automatic Capture Assessment Study
Brief Title: ULTRA Study for Pacemaker Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-CA-051205-B
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2007-07

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

INTERVENTIONS:
Device: Pacemaker with Automatic Capture

SUMMARY:
The ULTRA study will assess the difference in average ventricular voltage output for pacemaker patients randomized to Automatic Capture feature ON versus patients randomized to Automatic Capture feature OFF.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet current INSIGNIA® Ultra pacemaker indications
* Patients who will be programmed to a pacing mode of DDD, DDDR, VVI, VVIR, or VDD at the time of implant
* Patients who sign and date a Patient Informed Consent form at or prior to the implant visit
* Patients who remain in the clinical care of the enrolling physician in approved centers

Exclusion Criteria:

* Patients who will receive a single chamber device with an atrial lead only
* Patients who have chronic leads with a ventricular threshold of more than 4.0 V
* Patients whose life expectancy is less than 12 months
* Patients who are expected to receive a heart transplant during the duration of the study
* Patients who have or who are likely to receive a tricuspid valve prosthesis
* Patients who are currently enrolled in another investigational study that would directly impact the treatment or outcome of the ULTRA study.
* Patients who are younger than 18 years of age
* Patients who are pregnant
* Patients who are mentally incompetent and cannot sign a Patient Informed Consent form or comply with the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 950
Dates: Start 2005-07; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Average ventricular voltage output over time for patients randomized to Automatic Capture feature ON versus patients randomized to Automatic Capture feature OFF

SECONDARY OUTCOMES:
Compare automatic and manual threshold tests
Project device longevity

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Koplan, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Choi HY, Noh YH, Jin SJ, Kim YH, Kim MJ, Sung H, Jang SB, Lee SJ, Bae KS, Lim HS. Bioavailability and tolerability of combination treatment with revaprazan 200 mg + itopride 150 mg: a randomized crossover study in healthy male Korean volunteers. Clin Ther. 2012 Sep;34(9):1999-2010. doi: 10.1016/j.clinthera.2012.07.004. Epub 2012 Aug 1. PMID 22858177